CLINICAL TRIAL: NCT02272842
Title: The Effect of Vitamin B12 Supplementation in Nepali Infants on Growth and Development
Brief Title: Vitamin B12, Neurodevelopment and Growth in Nepal
Acronym: BeLive
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre For International Health (Other)
Collaborators: Tribhuvan University, Nepal (Other); NORCE Norwegian Research Centre AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 808734; U1111-1161-5187 (Other: WHO)
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-07

CONDITIONS: Development; Vitamin Deficiency; Malnutrition
Keywords: Nepal; Cobalamin; Neurodevelopment; Stunting; Growth
MeSH Terms: conditions — Avitaminosis; Malnutrition; Growth Disorders | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin B12 (Experimental): A paste containing vitamin B12 2µg per 10 mL administered every day. The paste also contains 1 RDA of several other vitamins. The paste is produced by Compact (Norway / India)
  Interventions: Dietary Supplement: Vitamin B12
- Placebo (Placebo Comparator): A paste containing no vitamin administered every day. The paste also contains 1 RDA of several vitamins, but no vitamin B12. The paste is produced by Compact (Norway / India)
  Interventions: Dietary Supplement: Vitamin B12

INTERVENTIONS:
Dietary Supplement: Vitamin B12 — Vitamin B12 in a multivitamin paste.
  Other Names: Cobalamin

SUMMARY:
Rationale: Globally, vitamin B12 deficiency is one of the most common micronutrient deficiencies. The only relevant source of Vitamin B12 is animal-source foods. Vitamin B12 is crucial for normal cell division and is necessary for brain growth as well as for the maintenance of its normal function. Deficiency is also associated with impaired growth. In a previous study, we demonstrated that vitamin B12 administration over a period of six months enhanced growth, and scores on a neuro-developmental test in young Indian children. However, the overall effect was small and, for the developmental scores significant only in those that were malnourished at the start of the study.

Our findings need to be verified in trials targeting younger, malnourished children and with longer supplementation time.

Hypothesis: This proposed study will test three hypotheses; to measure to what extent 2 recommended daily allowances (RDA) of vitamin B12 administration for one year to stunted children improves; 1) growth, 2) neurodevelopment, and 3) hemoglobin concentration.

Study design: Randomized placebo-controlled trial. Half of the children will receive a paste containing vitamin B12, the other half the same paste but without vitamin B12.

Study participants and site: 600 malnourished infants in Bhaktapur municipality in Nepal. In this population we have demonstrated that vitamin B12 deficiency and poor growth is common in early childhood.

Intervention: Daily administration of a paste containing vitamin B12 or placebo for 12 months

Data: The main outcomes of this study are scores on developmental assessments tools and growth measured every month for 12 months.

DETAILED DESCRIPTION:
Scientific basis: Globally, vitamin B12 deficiency is one of the most common micronutrient deficiencies. The only relevant source of vitamin B12 is animal-source foods. Vitamin B12 is crucial for normal cell division and differentiation and is necessary for the development and initial myelination of the central nervous system as well as for the maintenance of its normal function. Deficiency is also associated with impaired infant and child growth.

In a previous clinical trial, we demonstrated that vitamin B12 administration over a period of six months enhanced growth and neurodevelopment in young Indian children. The overall effect on growth was significant but small. We saw an effect on both ponderal (weight for age z scores) and linear (height for age z scores) growth. However, the overall effects were driven by the effects in the subgroups of children who were wasted, underweight or stunted at baseline, and no effect in the children who were not malnourished at baseline. This effect modification was significant for all three (stunting, wasting, and underweight) baseline variables. Similarly, the effect of the intervention on neurodevelopmental scores was also strongest in the subgroup of children that were stunted.

We have for the last 15 years undertaken studies on dietary intake and status in women and children in Bhaktapur, Nepal. In this site, vitamin B12 deficiency is very common. The objective of the proposed study is to measure to what extent administration of 2 RDA of vitamin B12 to stunted children from the last half of infancy and for 12 months affect neurodevelopment, growth and hemoglobin concentration.

Hypothesis: Daily supplementation of 2 RDA of vitamin B12 in young Nepali children for 12 months improves neurodevelopment, growth and hemoglobin concentration.

Study design: Individually randomized placebo controlled, double blind trial. Children will be identified in the community and stunted children will be randomized to daily receive a paste containing vitamin B12 or a placebo paste. The paste will be delivered by trained field workers every day and by the caregivers on Saturdays and public holidays.

Study participants and site: 600 stunted children aged 6 to 11 months in Bhaktapur municipality and surrounding areas.

Intervention: Daily administration of a paste containing vitamin B12 or placebo for 12 months.

Comparator: Placebo, identical to the vitamin B12 supplements.

Data: Primary outcomes: (i) neurodevelopmental scores measured by Bayley Scales of Infant and Toddler Development 3rd edition and the Ages and Stages Questionnaire 3rd edition after 6 and 12 months of supplementation (ii) growth measured by change in height for age, weight for age and weight for height z-score from study start to end study and growth velocity z scores during the six first and six last months of supplementation (iii) hemoglobin concentration after 12 months of supplementation. Secondary: (i) cognitive development in children measured approximately 3 and 6 years after enrollment, (ii) linear and ponderal growth measured 2 and 3 years after enrollment, (iii) hemoglobin concentration measured 2 and 3 years after enrollment. All secondary outcomes require additional funding.

Relevance for programs and public health: Improved learning ability and growth in young malnourished children. If the supplementation is effective this will have consequences for dietary recommendation to malnourished children worldwide. In contrast to most other relevant nutritional interventions, vitamin B12 is inexpensive and our body has the ability to store vitamin B12, up to years. Thus, improving the status of this nutrient for a limited time period may have impact on learning and productivity beyond the time of administration and help to lift poor children out of the vicious cycle of poverty and malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 11 months
* Stunted
* Availability of informed verbal consent
* Plan to reside in the area for the next 12 months

Exclusion Criteria:

* Severe systemic illness requiring hospitalization
* Severe malnutrition, i.e. weight for height < -3 z of the WHO standard for this age group. For ethical reasons these children require micronutrient supplementation and adequate medical care.
* Lack of consent
* Taking B vitamin supplements that include vitamin B12.
* Severe anemia (Hb < 7 g/dL). This would be a temporary exclusion and the children will be enrolled if they are successfully treated.
* Ongoing acute infection with fever or infection that requires medical treatment. This would be a temporary exclusion and the children will be enrolled after recovery.

Ages: 6 Months to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2024-12-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Prakash S Shrestha, MD, Principal Investigator — Tribhuvan University, Nepal; Tor A Strand, MD/PhD, Principal Investigator — Innlandet Hospital Trust / University of Bergen
Locations (1):
- Siddhi Memorial Hospital (SMH),Bhelukhel, Bhimsensthan, Bhaktapur, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Data available on request. In order to meet ethical requirements for the use of confidential patient data, requests must be approved by the Nepal Health Research Council (NHRC) and the Regional Committee for Medical and Health Research Ethics in Norway. Requests for data should be sent to the authors, by contacting NHRC (http://nhrc.gov.np), or by contacting the Department of Global Health and Primary Care at the University of Bergen (post@igs.uib.no).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon publication of the main outcomes.
Access Criteria: The protocols and the plan of analyses will be available with the main publication. IPD will be available following an application process which involves the ethical committees in Norway and Nepal

REFERENCES:
- [Background] Taneja S, Strand TA, Kumar T, Mahesh M, Mohan S, Manger MS, Refsum H, Yajnik CS, Bhandari N. Folic acid and vitamin B-12 supplementation and common infections in 6-30-mo-old children in India: a randomized placebo-controlled trial. Am J Clin Nutr. 2013 Sep;98(3):731-7. doi: 10.3945/ajcn.113.059592. Epub 2013 Jul 31. PMID 23902779
- [Background] Strand TA, Taneja S, Ueland PM, Refsum H, Bahl R, Schneede J, Sommerfelt H, Bhandari N. Cobalamin and folate status predicts mental development scores in North Indian children 12-18 mo of age. Am J Clin Nutr. 2013 Feb;97(2):310-7. doi: 10.3945/ajcn.111.032268. Epub 2013 Jan 2. PMID 23283502
- [Background] Black MM. Effects of vitamin B12 and folate deficiency on brain development in children. Food Nutr Bull. 2008 Jun;29(2 Suppl):S126-31. doi: 10.1177/15648265080292S117. PMID 18709887
- [Background] Black MM. Micronutrient deficiencies and cognitive functioning. J Nutr. 2003 Nov;133(11 Suppl 2):3927S-3931S. doi: 10.1093/jn/133.11.3927S. PMID 14672291
- [Derived] Ulak M, Kvestad I, Chandyo RK, Schwinger C, Basnet S, Shrestha M, Ranjitkar S, Nguyen LV, Corona-Perez D, De Vivo I, Ueland PM, McCann A, Strand TA. The Effect of Vitamin B12 Supplementation on Leukocyte Telomere Length in Mildly Stunted Nepalese Children: A Secondary Outcome of a Randomized Controlled Trial. J Nutr. 2024 Aug;154(8):2543-2550. doi: 10.1016/j.tjnut.2023.10.015. Epub 2023 Oct 31. PMID 37918674
- [Derived] Chandyo RK, Schwinger C, Kvestad I, Ulak M, Ranjitkar S, Shrestha M, Nguyen LV, Corona-Perez D, DeVivo I, Shrestha L, Strand TA. The association between household biomass fuel use and leukocyte telomere length among toddlers in Bhaktapur, Nepal. J Expo Sci Environ Epidemiol. 2023 May;33(3):448-454. doi: 10.1038/s41370-022-00474-1. Epub 2022 Sep 22. PMID 36138138
- [Derived] Hysing M, Strand TA, Chandyo RK, Ulak M, Ranjitkar S, Schwinger C, Shrestha M, Kvestad I. The effect of vitamin B12-supplementation on actigraphy measured sleep pattern; a randomized control trial. Clin Nutr. 2022 Feb;41(2):307-312. doi: 10.1016/j.clnu.2021.11.040. Epub 2021 Dec 6. PMID 34999324
- [Derived] Strand TA, Ulak M, Hysing M, Ranjitkar S, Kvestad I, Shrestha M, Ueland PM, McCann A, Shrestha PS, Shrestha LS, Chandyo RK. Effects of vitamin B12 supplementation on neurodevelopment and growth in Nepalese Infants: A randomized controlled trial. PLoS Med. 2020 Dec 1;17(12):e1003430. doi: 10.1371/journal.pmed.1003430. eCollection 2020 Dec. PMID 33259482
- [Derived] Strand TA, Ulak M, Chandyo RK, Kvestad I, Hysing M, Shrestha M, Basnet S, Ranjitkar S, Shrestha L, Shrestha PS. The effect of vitamin B12 supplementation in Nepalese infants on growth and development: study protocol for a randomized controlled trial. Trials. 2017 Apr 21;18(1):187. doi: 10.1186/s13063-017-1937-0. PMID 28431557
- See also: Link to the founding source. — https://www.thrasherresearch.org/SitePages/current-grants-all.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment commenced in April 2015 and ended in February 2017. All children were supplemented daily for one year. Follow-up ended in February 2018
Groups:
- Placebo: A paste containing no vitamin B12 administered every day. The paste also contains 1 RDA of several vitamins, but no vitamin B12. The paste is produced by Compact (Norway / India)
  Placebo B12: Placebo B12 in a multivitamin paste.
Period: Overall Study
Arm/Group | Vitamin B12 | Placebo
Started | 300 | 300
Completed | 284 | 290
Not Completed | 16 | 10
Not completed — Lost to Follow-up | 8 | 8
Not completed — Withdrawal by Subject | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin B12 | Placebo | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Continuous [Mean (Standard Deviation); unit: Months] | 8.0 (1.8) | 8.1 (1.8) | 8.0 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 142 | 291
  Male | 151 | 158 | 309
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Nepalese | 300 | 300 | 600
Length (cm) [Mean (Standard Deviation); unit: cm] | 65.837 (3.0) | 65.94 (2.9) | 65.9 (3.0)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 7.3 (0.92) | 7.3 (0.92) | 7.3 (.92)

OUTCOME MEASURES:

1. Primary Outcome: The Bayley Scales of Infant Development Version 3
Description: Cognitive, Fine Motor, Gross Motor, Receptive language, and Expressive language scaled scores of the Bayley Scales of Infant Development version 3. This scale measures different aspects of neurodevelopment. The mean (SD) scores are usually 100 (15), and 95% of the population has scores between 70 and 130 (theoretical max/means 0/200). The higher scores, the better neurodevelopment; the scale is normalized on age.
Time Frame: 12 months
Population: Cognitive, Fine Motor, Gross Motor, Receptive language, and Expressive language scaled scores of the Bayley Scales of Infant Development version 3. This scale measures different aspects of neurodevelopment. The mean (SD) scores are usually 100 (15), and 95% of the population has scores between 70 and 130 (theoretical max/means 0/200). The higher scores, the better neurodevelopment; the scale is normalized on age.
Measure: Mean (Standard Deviation); unit: Scaled Scores
Arm/Group | Vitamin B12 | Placebo
Number analyzed (Participants) | 289 | 283
Scaled Scores
  Cognitive | 8.1 (1.6) | 8.2 (1.5)
  Receptive language | 9.0 (2.3) | 8.9 (2.5)
  Expressive language | 8.6 (2.6) | 8.5 (2.4)
  Fine Motor | 10.7 (1.6) | 10.9 (1.8)
  Gross Motor | 9.2 (2.0) | 9.1 (1.7)
Statistical Analysis 1: Comparison: Vitamin B12 vs Placebo; Test type: Superiority — The study had 80% power to detect a standardized effect size of 0.22 and had 90% power to detect an effect size of 0.28. In these calculations, we assumed a loss to follow-up of 10%. Details on the samples size calculations are also presented in the previously published protocol paper; p > .16, t-test, 2 sided — The main analysis was the change in cognitive scores from baseline until the end of the intervention; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-.54 to .87], Standard Error of Mean .35 — This is the P-value for the effect on the cognitive scores

2. Primary Outcome: Hemoglobin Concentration
Description: Change in hemoglobin concentration from baseline to end study.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Vitamin B12 | Placebo
Number analyzed (Participants) | 288 | 281
g/dl | 1.1 (1.1) | 1.0 (1.2)

3. Secondary Outcome: Growth Velocity Over the First Six Months of Supplementation
Description: length and weight growth velocity z scores during supplementation z-scores, growth velocity. theoretical values -10 to 10 The higher the value, the faster the growth.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2025-01

4. Secondary Outcome: Predictors for Neurodevelopment in Young Nepali Children
Description: Using the collected data, identify morbidity, stimulation, nutrition, socioeconomic related predictors for neurodevelopment.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2024-01

5. Secondary Outcome: Identify Subgroups of Children Who Benefit From Vitamin B12 Supplementation
Description: Based on selected baseline variables we will identify subgroups who benefit from vitamin B12 supplementation
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2025-01

6. Secondary Outcome: The Effect of Vitamin B12 Supplementation on Markers of Vitamin B Status
Description: We will draw a blood sample at study start and at end study to measure to what extent vitamin status is altered.
Time Frame: 12 months
Population: Comparing mean plasma concentration of cobalamin between the study groups.
Measure: Mean (Standard Deviation); unit: mol/L
Arm/Group | Vitamin B12 | Placebo
Number analyzed (Participants) | 277 | 286
mol/L
  Cobalamin | 316.3 (1.7) | 290.1 (1.6)
  homocysteine' | 6.6 (1.3) | 8.2 (1.4)
  Methyl Malonic acid | 0.3 (1.9) | .4 (2.1)

7. Secondary Outcome: Neurodevelopment Measured by Other Tools.
Description: We will measure to what extent vitamin B12 supplementation improves neurodevelopment measured by other tools such as the Ages and Stages Questionnaire (version 3) and the NEPSY II test.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2024-01

8. Secondary Outcome: Immediate Adverse Effects of the Intervention
Description: We will investigate side effects such as pain, nausea, vomiting, regurgitation, allergic reactions and others after each dose of the intervention.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin B12 | Placebo
Number analyzed (Participants) | 26 | 17
Participants
  Urinary tract infections | 3 | 0
  Lower respiratory infections | 8 | 10
  Seizure related illness | 7 | 2
  Constipation | 1 | 1
  Other (surgical, diarrhea, sepsis, etc.) | 7 | 4

9. Secondary Outcome: Leucocyte Telomere Length
Description: Relative leucocyte telomere length at end of the study period. Estimated by real-time PCR analysis
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2024-01

10. Secondary Outcome: Sleep Duration
Description: Using actigraph and a structured questionaire on all children at baseline and at end of study measure the extent to which the intervention affects sleep.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2025-02

11. Other Pre Specified Outcome: Extended Followup: Neurodevelopment (IQ)
Description: Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition. This is a test of general abilities ("IQ-test") Expected mean (SD): 100 (15), higher value indicate better cognitive functioning. Range approx. 40-140
Time Frame: 3 years
Population: All children who were available for assessment
Measure: Mean (Standard Deviation); unit: IQ points
Arm/Group | Vitamin B12 | Placebo
Number analyzed (Participants) | 269 | 264
IQ points | 84.4 (8.4) | 85.0 (8.6)
Statistical Analysis 1: Comparison: Vitamin B12 vs Placebo; Comparing mean differences between the two study arms; Test type: Superiority — the means were compared using Students t-test; p > .3, t-test, 2 sided — Mean difference -0.5 points in the Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition. 95 % Confidence Interval of the mean difference: (-1.97, 0.94); Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.97 to 0.94]

12. Other Pre Specified Outcome: Surrogate Markers for Neurodevelopment
Description: If funding allows, measure other markers related to neurodevelopment such as Brain Derived Neurotrophic Factor
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2024-01

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Vitamin B12 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/300
Serious Adverse Events (participants affected / at risk) | 2/300 | 0/300
Other Adverse Events (participants affected / at risk) | 70/300 | 63/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin B12 (N=300) | Placebo (N=300)
Abscess (Infections and infestations) | 1 (1) | 0 (0) — admitted with diagnosis of abscess over left lateral neck (staph aureus isolated) treated : inj flucloxacillin and inj cefotaxime
Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The child was burn with hot water on face and head admitted to a tertiary hosptial
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin B12 (N=300) | Placebo (N=300)
Regurgitation following paste administration. (Gastrointestinal disorders) | 70 (141) | 63 (134)
Urinary tract infection (Renal and urinary disorders) | 3 (3) | 0 (0)
Lower respiratory infection (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 8 (10)
Febrile seizures (Nervous system disorders) | 6 (7) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT02272842/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT02272842/SAP_001.pdf